CLINICAL TRIAL: NCT03797222
Title: Vitamin E Supplementation in Hyperinsulinism/Hyperammonemia Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elizabeth A Rosenfeld (Other)
Collaborators: University of Pennsylvania (Other); Lawson Wilkins Pediatric Endocrine Society (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Elizabeth A Rosenfeld, Attending Physician, Children's Hospital of Philadelphia
Organization: Children's Hospital of Philadelphia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17-014550; T32DK063688 (NIH)
Record Dates: First submitted 2019-01-06; First posted 2019-01-09 (Actual); Results first posted 2022-11-25 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Hyperinsulinism-Hyperammonemia Syndrome
Keywords: hyperinsulinism; hyperammonemia; hypoglycemia; vitamin e
MeSH Terms: conditions — Hyperinsulinemic hypoglycemia, familial, 6; Hyperinsulinism; Hyperammonemia; Hypoglycemia | interventions — Vitamin E; alpha-Tocopherol

STUDY DESIGN:
Intervention Model Description: This open-label tolerability and feasibility pilot clinical study will use a before-and-after design, with blood tests and fasting oral protein tolerance test performed prior to and after 2 weeks of daily oral Vitamin E supplementation in individuals with HI/HA syndrome.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vitamin E Supplementation (Experimental): Daily oral supplementation with Vitamin E (alpha-tocopherol) for 2 weeks.
  Interventions: Dietary Supplement: Vitamin E

INTERVENTIONS:
Dietary Supplement: Vitamin E — Subjects will take an oral Vitamin E (alpha-tocopherol) supplement once daily with a fat-containing meal for 2 weeks. The dose will be based on subject age (150 IU if 1-3 years old, 300 IU if 4-8 years old, 450 IU if 9-17 years old, 600 IU if >17 years old). Formulations include 50 IU/mL liquid and 200 IU capsules. The liquid formulation will be used for subjects who will receive <600 IU daily, or for any subjects who prefer liquid medication to capsules.
  Other Names: alpha-tocopherol

SUMMARY:
Investigators will assess the tolerability of oral Vitamin E supplementation in subjects with congenital hyperinsulinism (HI) and hyperammonemia (HA) syndrome.

DETAILED DESCRIPTION:
Congenital hyperinsulinism (HI) is a rare disorder of pancreatic beta cell insulin secretion that causes persistent and severe hypoglycemia starting at birth. Hyperinsulinism/hyperammonemia (HI/HA) syndrome is the second most common type of congenital HI and is caused by activating mutations in glutamate dehydrogenase (GDH). Patients with HI/HA exhibit fasting hyperinsulinemic hypoglycemia, protein-induced hypoglycemia, hyperammonemia, seizures, and intellectual disability independent of hypoglycemia. These effects result from abnormal GDH activity in the beta cells, liver and kidney cells, neurons, and astrocytes. The only available treatment for HI/HA syndrome is diazoxide, which acts on the beta cells to decrease insulin secretion but has no effect on GDH activity itself or on other cell types. Thus, there remains a significant unmet need for improved therapies for this disorder. Preliminary data show that Vitamin E (alpha-tocopherol) inhibits GDH activity in cell lines and improves hypoglycemia in a GDH HI mouse model. Based on these preclinical studies, Investigators hypothesize that Vitamin E will inhibit GDH activity and may impact hyperinsulinemic hypoglycemia and hyperammonemia in subjects with HI/HA syndrome. This hypothesis will be tested in a future study. In this initial pilot study, investigators will assess the tolerability of oral Vitamin E supplementation in subjects with HI/HA syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Individuals age ≥12 months and ≤40 years
* Diagnosis of HI/HA syndrome
* On diazoxide therapy for treatment of hypoglycemia
* Females ≥11 years of age or menstruating must have a negative urine/serum pregnancy test and must use an acceptable method of contraception, including abstinence, a barrier method (diaphragm or condom), Depo-Provera, or an oral contraceptive, for the duration of the study.
* Informed consent for participants ≥18 years. Parental/guardian permission (informed consent) and, if appropriate, child assent for participants <18 years.

Exclusion Criteria:

* Individuals age <12 months or >40 years
* Individuals who have experienced an allergic reaction to Vitamin E
* Individuals with a known allergy to dairy, whey, or soy
* On concurrent therapy with a medication known to be metabolized by the CYP3A pathway
* Individuals with a known increased risk of bleeding (bleeding disorder or on antiplatelet or anticoagulation therapy)
* Vitamin E supplementation within 30 days prior to enrollment, including multivitamins containing Vitamin E
* Severe hypoglycemia (plasma glucose <50 mg/dL on repeat checks using home glucose meter) more than once weekly within 30 days prior to enrollment.
* Evidence of a medical condition that might alter results or compromise the interpretation of results, including active infection, kidney failure, severe liver dysfunction, severe respiratory or cardiac failure.
* Evidence of severe hematologic abnormality including severe anemia and/or thrombocytopenia.
* Any investigational drug use within 30 days prior to enrollment.
* Pregnant or lactating females.
* Parents/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.
* Unable to provide informed consent (e.g. impaired cognition or judgment).
* Parents/guardians or subjects with limited English proficiency.

Ages: 1 Year to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Rosenfeld, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palladino AA, Stanley CA. The hyperinsulinism/hyperammonemia syndrome. Rev Endocr Metab Disord. 2010 Sep;11(3):171-8. doi: 10.1007/s11154-010-9146-0. PMID 20936362
- [Background] Snider KE, Becker S, Boyajian L, Shyng SL, MacMullen C, Hughes N, Ganapathy K, Bhatti T, Stanley CA, Ganguly A. Genotype and phenotype correlations in 417 children with congenital hyperinsulinism. J Clin Endocrinol Metab. 2013 Feb;98(2):E355-63. doi: 10.1210/jc.2012-2169. Epub 2012 Dec 28. PMID 23275527
- [Background] Hsu BY, Kelly A, Thornton PS, Greenberg CR, Dilling LA, Stanley CA. Protein-sensitive and fasting hypoglycemia in children with the hyperinsulinism/hyperammonemia syndrome. J Pediatr. 2001 Mar;138(3):383-9. doi: 10.1067/mpd.2001.111818. PMID 11241047
- [Background] Stanley CA, Baker L. Hyperinsulinism in infancy: diagnosis by demonstration of abnormal response to fasting hypoglycemia. Pediatrics. 1976 May;57(5):702-11. PMID 940710
- [Background] Li M, Smith CJ, Walker MT, Smith TJ. Novel inhibitors complexed with glutamate dehydrogenase: allosteric regulation by control of protein dynamics. J Biol Chem. 2009 Aug 21;284(34):22988-3000. doi: 10.1074/jbc.M109.020222. Epub 2009 Jun 15. PMID 19531491
- [Background] McBurney MI, Yu EA, Ciappio ED, Bird JK, Eggersdorfer M, Mehta S. Suboptimal Serum alpha-Tocopherol Concentrations Observed among Younger Adults and Those Depending Exclusively upon Food Sources, NHANES 2003-20061-3. PLoS One. 2015 Aug 19;10(8):e0135510. doi: 10.1371/journal.pone.0135510. eCollection 2015. PMID 26287975
- [Background] Ulatowski L, Manor D. Vitamin E trafficking in neurologic health and disease. Annu Rev Nutr. 2013;33:87-103. doi: 10.1146/annurev-nutr-071812-161252. Epub 2013 Apr 29. PMID 23642196
- [Background] Pfeiffer CM, Sternberg MR, Schleicher RL, Haynes BM, Rybak ME, Pirkle JL. The CDC's Second National Report on Biochemical Indicators of Diet and Nutrition in the U.S. Population is a valuable tool for researchers and policy makers. J Nutr. 2013 Jun;143(6):938S-47S. doi: 10.3945/jn.112.172858. Epub 2013 Apr 17. PMID 23596164
- [Background] Ferslew KE, Acuff RV, Daigneault EA, Woolley TW, Stanton PE Jr. Pharmacokinetics and bioavailability of the RRR and all racemic stereoisomers of alpha-tocopherol in humans after single oral administration. J Clin Pharmacol. 1993 Jan;33(1):84-8. doi: 10.1002/j.1552-4604.1993.tb03909.x. PMID 8429120
- [Background] Treberg JR, Clow KA, Greene KA, Brosnan ME, Brosnan JT. Systemic activation of glutamate dehydrogenase increases renal ammoniagenesis: implications for the hyperinsulinism/hyperammonemia syndrome. Am J Physiol Endocrinol Metab. 2010 Jun;298(6):E1219-25. doi: 10.1152/ajpendo.00028.2010. Epub 2010 Mar 23. PMID 20332361

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vitamin E Supplementation
Started | 14
Completed | 13
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Vitamin E Supplementation
Number analyzed (Participants) | 14
Age, Continuous [Median (Full Range); unit: years] | 8 [2 to 28]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 6
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Tolerability of Vitamin E Based on Responses to a Subject/Parent-reported Symptom Questionnaire After Vitamin E Supplementation Compared to Baseline
Description: The following symptoms will be scored as either "none" (did not occur)=0, "mild" (minimal symptoms, no treatment needed)=1, "moderate" (symptoms requiring treatment at home or as an outpatient=2, or "severe" (symptoms requiring hospitalization or emergency room visit, or life-threatening or potentially life-threatening symptoms)=4:
  Seizure, Headache, Vision change/blurred vision, Weakness, Fatigue, Nausea, Vomiting, Diarrhea, Stomach pain, Constipation, Bruising, Bleeding, Rash, Itching, Other
  Symptom scores will be summed to yield a Tolerability Questionnaire Score for each participant. The Tolerability Questionnaire Score has a minimum score of 0 (symptoms did not occur) and a maximum score of 60 (all of the measured symptoms occurred, each with severe designation).
  The number (count) of participants with an increase in Tolerability Questionnaire Score from baseline to 2 weeks (following Vitamin E supplementation) will be reported.
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin E Supplementation
Number analyzed (Participants) | 13
Participants | 2

2. Secondary Outcome: Plasma Alpha-tocopherol Concentration
Description: change in fasting plasma alpha-tocopherol concentration following Vitamin E supplementation (2 weeks [visit 2] - baseline [visit 1])
Time Frame: 2 weeks
Population: The 2 week (visit 2) laboratory draw was unable to be obtained for 1 participant, yielding n=12 analyzed for this outcome
Measure: Mean (Standard Deviation); unit: micromolar
Arm/Group | Vitamin E Supplementation
Number analyzed (Participants) | 12
micromolar | 18.6 (12.5)

3. Secondary Outcome: Delta-plasma Glucose Concentration
Description: change in delta-glucose concentration (fasting plasma glucose - nadir plasma glucose during oral protein tolerance test) following Vitamin E supplementation (2 weeks [visit 2] - baseline [visit 1])
Time Frame: 2 weeks
Population: Per the study protocol, the oral protein tolerance test was not repeated at 2 weeks (visit 2) if the baseline (visit 1) oral protein tolerance test was not tolerated. Of the 13 participants who completed the study, 7 did not tolerate the baseline (visit 1) oral protein tolerance test. The 2 week (visit 2) oral protein tolerance test was performed in 6 participants. Oral protein tolerance test parameters were analyzed for these 6 participants.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Vitamin E Supplementation
Number analyzed (Participants) | 6
mg/dL | 1.1 (8.3)

4. Secondary Outcome: Fasting Plasma Glucose Concentration
Description: change in fasting plasma glucose concentration following Vitamin E supplementation (2 weeks [visit 2] - baseline [visit 1])
Time Frame: 2 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Vitamin E Supplementation
Number analyzed (Participants) | 12
mg/dL | -0.3 (6.5)

5. Secondary Outcome: Nadir Plasma Glucose Concentration
Description: change in nadir plasma glucose concentration during oral protein tolerance test following Vitamin E supplementation (2 weeks [visit 2] - baseline [visit 1])
Time Frame: 2 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Vitamin E Supplementation
Number analyzed (Participants) | 6
mg/dL | 0.01 (9.46)

6. Secondary Outcome: Fasting Plasma Insulin Concentration
Description: change in fasting plasma insulin concentration following Vitamin E supplementation (2 weeks [visit 2] - baseline [visit 1])
Time Frame: 2 weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: uIU/mL
Arm/Group | Vitamin E Supplementation
Number analyzed (Participants) | 12
uIU/mL | -2.4 (4.4)

7. Secondary Outcome: Peak Plasma Insulin Concentration
Description: change in peak plasma insulin concentration during oral protein tolerance test following Vitamin E supplementation (2 weeks [visit 2] - baseline [visit 1])
Time Frame: 2 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: uIU/mL
Arm/Group | Vitamin E Supplementation
Number analyzed (Participants) | 6
uIU/mL | -6.3 (18.2)

8. Secondary Outcome: Delta-plasma Insulin Concentration
Description: change in delta-plasma insulin concentration (peak plasma insulin - fasting plasma insulin during oral protein tolerance test) following Vitamin E supplementation (2 weeks [visit 2] - baseline [visit 1])
Time Frame: 2 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: uIU/mL
Arm/Group | Vitamin E Supplementation
Number analyzed (Participants) | 6
uIU/mL | -5.2 (16.5)

9. Secondary Outcome: Fasting Plasma Ammonia Concentration
Description: change in fasting plasma ammonia concentration following Vitamin E supplementation (2 weeks [visit 2] - baseline [visit 1])
Time Frame: 2 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: micromolar
Arm/Group | Vitamin E Supplementation
Number analyzed (Participants) | 12
micromolar | 1.0 (31.6)

10. Secondary Outcome: Delta-plasma Ammonia Concentration
Description: change in delta-plasma ammonia concentration (plasma ammonia at 60 minutes - fasting plasma ammonia during oral protein tolerance test) following Vitamin E supplementation (2 weeks [visit 2] - baseline [visit 1])
Time Frame: 2 weeks
Population: The 2 week (visit 2) plasma ammonia at 60 minutes was not obtained in 1 participant in whom the visit 2 oral protein tolerance test was performed, yielding n=5 for analysis of this outcome.
Measure: Mean (Standard Deviation); unit: micromolar
Arm/Group | Vitamin E Supplementation
Number analyzed (Participants) | 5
micromolar | -3.4 (15.5)

11. Secondary Outcome: Hypoglycemia Frequency
Description: change in frequency of hypoglycemia (plasma glucose <70 mg/dL) detected on home glucose meter following Vitamin E supplementation (2 weeks [visit 2] - baseline [visit 1])
Time Frame: 2 weeks
Population: Home glucose meter testing was not performed by 3 participants, yielding n=10 analyzed for this outcome.
Measure: Mean (Standard Deviation); unit: Hypoglycemia events
Arm/Group | Vitamin E Supplementation
Number analyzed (Participants) | 10
Hypoglycemia events | 0.6 (2.3)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the 2 week study period.
Groups:
- Vitamin E Supplementation (All Doses): Daily oral supplementation with Vitamin E (alpha-tocopherol) for 2 weeks.
  Vitamin E: Subjects will take an oral Vitamin E (alpha-tocopherol) supplement once daily with a fat-containing meal for 2 weeks. The dose will be based on subject age (150 IU if 1-3 years old, 300 IU if 4-8 years old, 450 IU if 9-17 years old, 600 IU if >17 years old). Formulations include 50 IU/mL liquid and 200 IU capsules. The liquid formulation will be used for subjects who will receive <600 IU daily, or for any subjects who prefer liquid medication to capsules.
- Vitamin E 150 IU: Daily oral supplementation with Vitamin E (alpha-tocopherol) 150 IU for 2 weeks.
- Vitamin E 300 IU: Daily oral supplementation with Vitamin E (alpha-tocopherol) 300 IU for 2 weeks.
- Vitamin E 450 IU: Daily oral supplementation with Vitamin E (alpha-tocopherol) 450 IU for 2 weeks.
- Vitamin E 600 IU: Daily oral supplementation with Vitamin E (alpha-tocopherol) 600 IU for 2 weeks.
Arm/Group | Vitamin E Supplementation (All Doses) | Vitamin E 150 IU | Vitamin E 300 IU | Vitamin E 450 IU | Vitamin E 600 IU
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/2 | 0/5 | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/2 | 0/5 | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 9/14 | 1/2 | 2/5 | 3/3 | 3/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Vitamin E Supplementation (All Doses) (N=14) | Vitamin E 150 IU (N=2) | Vitamin E 300 IU (N=5) | Vitamin E 450 IU (N=3) | Vitamin E 600 IU (N=4)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 5 (6) | 0 (0) | 0 (0) | 2 (2) | 3 (4)
Vomiting (Gastrointestinal disorders) | 4 (6) | 1 (1) | 0 (0) | 2 (3) | 1 (2)
Increased menstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 0/0 (0) | 0/0 (0) | 0/2 (0) | 1/3 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-11): https://cdn.clinicaltrials.gov/large-docs/22/NCT03797222/Prot_SAP_000.pdf